CLINICAL TRIAL: NCT00461279
Title: Attachment Security as Mediator and Moderator of Outcome in Major Depression Following Interpersonal Therapy and Cognitive Behavior Therapy
Brief Title: Attachment Security as Mediator and Moderator of Outcome in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Carolina McBride, Dr. Carolina McBride, C.Psych, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 165/2006
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Major Depression
Keywords: attachment; depression; IPT; CBT; pharmacotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy; Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Behavioral: Cognitive Behavior Therapy
- 2 (Other)
  Interventions: Behavioral: Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Reframing and understanding cognitions of depression
  Arms: 1
Behavioral: Interpersonal Psychotherapy — Established psychotherapy for depression
  Arms: 2

SUMMARY:
In this study, the focus is on an individual's attachment security and its relation to treatment outcome in Major Depression.Adult attachment reflects how one seeks psychological and physical proximity to others for security and protection in times of stress. Researchers typically define four types of attachment security: one secure and three insecure (preoccupied, dismissing, and fearful). Adults with Major Depressive Disorder (MDD) will be randomly assigned to either Interpersonal Psychotherapy (IPT) or to Cognitive Behavior Therapy (CBT). The expectation is that adults with avoidant attachment styles will respond better to CBT, and adults with preoccupied attachment styles will respond better to IPT. Also, in comparison to CBT, outcome in IPT is hypothesized to be more closely related to change in attachment.

DETAILED DESCRIPTION:
At the current rate of increase, Major Depression, it will be the 2nd most disabling condition in the world by 2020, behind heart disease. There are now a number of effective treatments for depression. However, a significant number of people either partially recover from their depression after a course of treatment, or do not recover at all. For example, between 30% and 50% of depressed individuals taking an antidepressant are partially or totally resistant to the treatment, and more than ½ of patients in psychotherapy never achieve full remission. The goal of treatment of major depression should always be full remission. Not achieving full remission from depression is problematic as lingering symptoms are a powerful predictor of relapse.

One problem may be in the type of treatment that is offered to the individual. We know little about which clients benefit from which type of treatments and which clients do poorly. One individual may respond better to one type of treatment, while another individual may respond better to another type of treatment. The accurate identification of how an individual's characteristics interact with the type of treatment offered will help us match patients to the best-suited treatment for them, so we can optimize outcome.

One characteristic that may be related to treatment outcome is adult attachment security. Adult attachment reflects how one seeks psychological and physical proximity to others for security and protection in times of stress. Researchers typically define four types of attachment security: one secure and three insecure (preoccupied, dismissing, and fearful). Secure adults have a good sense of self-worth and are comfortable with intimacy. Preoccupied adults have an exaggerated desire for closeness and a heightened concern about rejection. Dismissing adults deny the value of close relationships and instead value self-reliance. Finally, fearful adults have a very negative sense of self and avoid intimacy because they fear rejection. Secure attachment has been linked to positive interpersonal relationships and psychological health and insecure attachment has been linked to overall psychological distress.

In this study, I focus on attachment security and its relation to treatment outcome. Adults with Major Depressive Disorder (MDD) will be randomly assigned to either Interpersonal Psychotherapy (IPT) or to Cognitive Behavior Therapy (CBT). The expectation is that adults with avoidant attachment styles will respond better to CBT, and adults with preoccupied attachment styles will respond better to IPT. Also, in comparison to CBT, outcome in IPT is hypothesized to be more closely related to change in attachment.

The power of this study lies in its considered integration of three important issues at the forefront of mental health today: MDD, attachment, and treatment. MDD is a leading cause of disability worldwide and theoretically and empirically related to attachment. Attachment theory is a primary paradigm in the developmental, social/personality, and clinical literatures, and forms the theoretical cornerstone for IPT. IPT and CBT, while successful to a degree, fail or partially fail in many cases. Successful outcome in IPT depends on successfully improving a patient's attachment representations; this is not the case in CBT where change in depression is associated with change in cognition. The fact that these treatments represent contrasting approaches in the context of attachment, affords us a unique opportunity to investigate the relationships between attachment and treatment outcome for two distinct treatments, and investigate whether an individual's attachment security interacts with the type of treatment offered to yield a better response for one type of treatment versus another. This research could have a major impact on tailoring treatment to patient characteristics to optimize treatment for major depression.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* meet the criteria for DSM-IV diagnosis of MDD based on the Structured Interview for DSM-IV, Axis I disorders (SCID-I; First et al., 1995)
* score > 16 on the 17-item HRSD (Hamilton, 1960).

Exclusion Criteria:

* Bipolar Disorder
* Schizoaffective Disorder
* Schizophrenia
* Substance Abuse
* Borderline or Antisocial Personality Disorder
* Organic Brain Syndrome
* ECT within the past 6 months
* concurrent active medical illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2006-08; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
HAMD | baseline and completion
BDI | baseline and completion

CONTACTS AND LOCATIONS:
Overall Officials: Carolina McBride, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research